CLINICAL TRIAL: NCT06435260
Title: To Explore the Efficacy of Hypofractionated Radiotherapy Followed by AG Regimen Chemotherapy Plus Camrelizumab Immunotherapy as Neoadjuvant Therapy for Borderline Resectable/Locally Advanced Pancreatic Cancer
Brief Title: Hypofractionated Radiotherapy +Chemotherapy+ Camrelizumab as Neoadjuvant Therapy for Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARK-pancreatic-001
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypofractionated radiotherapy+Camrelizumab+chemotherapy (Experimental): The patients with Borderline Resectable/locally advanced pancreatic cancer were treated with hypofractionated radiotherapy using the CyberKnife radiotherapy machine, which was as follows: PGTV=30Gy/5F(PTV≥25Gy/5F), 1 day, a total of 5 days; Chemotherapy combined with ICIs was started 5-7 days after the end of radiotherapy. The chemotherapy regimen was AG regimen (albumin paclitaxel 125mg/m2 d1,8 + gemcitabine 1000mg/m2 d1,8 q3w). The ICIs regimen consisted of 4 cycles of camrelizumab 200mg q21d (on the first day of each cycle). The efficacy was evaluated within 2 weeks after the end of the above-mentioned neoadjuvant therapy, and surgical treatment was performed for patients who were evaluated as operable and those who had a clear willingness to undergo surgery. After surgery, adjuvant chemotherapy and ICIs of the original scheme were determined according to the patient's tolerance and independent willingness, and then the clinical follow-up period was entered.
  Interventions: Drug: Camrelizumab+chemotherapy; Radiation: hypofractionated radiotherapy

INTERVENTIONS:
Drug: Camrelizumab+chemotherapy — Chemotherapy combined with ICIs was started 5-7 days after the completion of radiotherapy:
  AG: intravenous nab-paclitaxel 125 mg/m2 and gemcitabine 1000mg/m2 d1,8, q3w, 4 cycles.
  Camrelizumab: 200mg, iv, 30min, q3w, 4 cycles.
Radiation: hypofractionated radiotherapy — Hypofractionated radiotherapy:PGTV=30Gy/5F(PTV≥25Gy/5F),

SUMMARY:
The purpose of this study is to assess surgical conversion rate and the immediate and long-term outcomes to patients who receive hypofractionated radiotherapy and AG combined with camrelizumab immunotherapy of Borderline Resectable/locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 to 75 years old, male or female;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
3. Tumor was located in the pancreas;
4. Pathological diagnosis was pancreatic ductal adenocarcinoma or acinar cell carcinoma;
5. No distant metastasis;
6. The pancreatic tumor is located more than 1cm away from the duodenum；
7. Clinical assessment was locally advanced or critical for resectable.

Locally advanced pancreatic cancer diagnostic criteria: (1) due to tumor invasion, venous occlusion or involving a wide range of superior mesenteric vein branch of jejunum, cannot safely - superior mesenteric vein reconstruction. ② (pancreatic head/uncinate process tumors) tumor contact with superior mesenteric artery or celiac artery > 180°. Tumor contact with superior mesenteric artery or coeliac trunk artery > 180°, tumor contact with coeliac trunk artery and invasion of abdominal aorta.

Critical for resectable pancreatic cancer diagnostic criteria: (1) contact with portal vein tumor - superior mesenteric vein > 180 °, 180 ° or less or contact combined intravenous contour irregular or venous thrombosis, but safety is complete resection and reconstruction; The tumor contacted the inferior vena cava. ② (pancreatic head/uncinate process tumors) the tumors contacting the common hepatic artery, but not involving the celiac artery or the origin of the left and right hepatic arteries, can be completely resected and safely reconstructed; Superior mesenteric artery tumor contact 180 ° or less; The tumor contacts the aberrant arteries (such as accessory right hepatic artery, alternative right hepatic artery, alternative common hepatic artery, etc.). (pancreatic body and tail tumors) tumor contact with superior mesenteric artery ≤180°; Tumor contact with celiac artery ≤180°; 7.There was no history of immune system diseases, other malignant tumors, myocarditis, coronary heart disease, other cardiovascular and cerebrovascular diseases, thyroid dysfunction, liver and kidney diseases, psychiatric diseases, infectious diseases, or systemic diseases other than those mentioned above.

Participants were willing to join in this study, good adherence and written informed consent.

Exclusion Criteria:

1. Patients who did not meet these inclusion criteria;
2. Poor cognitive ability, inability to answer questions, inability to fill out questionnaires, or mental disorders;
3. The investigators think inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
a.R0-resection rate | One week after surgery
  The tumor was completely removed during surgery, and the cutting margins were also negative when viewed microscopically

SECONDARY OUTCOMES:
Surgical conversion rate | 2 to 4 weeks after neoadjuvant therapy
  Tumors that were otherwise unresectable were transformed into surgically resectable tumors.
Tumor regression rate | One week after surgery
  Degree of tumor response to neoadjuvant therapy
Objective response rate (ORR) | through study completion，an average of 3 year
  It refers to the proportion of patients who achieve a prespecified reduction in tumor volume (CR/PR) and maintain the minimum time requirements according to accepted response evaluation criteria (e.g., RECIST in solid tumors, version 1.1).
Disease control rate (DCR) | through study completion，an average of 3 year
  It refers to the proportion of patients who achieve a prespecified reduction in tumor volume (CR/PR/SD) and maintain the minimum time requirements according to accepted response evaluation criteria (e.g., RECIST in solid tumors, version 1.1).
3-year Overall survival (OS) | Three years from enrollment
  The time between the start of randomization and death from any cause
3-year Event Free Survival (EFS) | Three years from enrollment
  The time from randomization until disease progression, treatment discontinuation for any cause, or death.
Adverse events | From enrollment to the end of treatment at 8 weeks
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. The number of participants with adverse events will be recorded at each treatment visit.
Quality of life scores | 1 years after therapy
  Evaluate the quality of life according to The World Health Organization quality of life (WHOQOL) -BREF. The minimum value is 1, the maximum value is 5. And higher scores mean a better outcome. The number of participants with quality of life will be recorded at each treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Li Peng, Principal Investigator — Fourth Hospital of Hebei Medical; Fengpeng Wu, Principal Investigator — Fourth Hospital of Hebei Medical
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No